CLINICAL TRIAL: NCT05765513
Title: Intra-pocket Injection of a Freshly Manufactured 35 kDa Hyaluronan Fragment HA35 Reduces the Gingival Discomfort as Well as Gingival Redness and Bleeding of Patients With Periodontitis: A Clinical Study
Brief Title: HA35 Treatment the Gingival Discomfort as Well as Gingival Redness and Bleeding of Patients With Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dove Medical Press Ltd (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: hui20050910
Record Dates: First submitted 2023-02-22; First posted 2023-03-13 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-02

CONDITIONS: Periodontitis
Keywords: 35 kDa low molecular hyaluronan fragment; HA35; Tissue permeability; Intra-pocket injection; Gingival redness and bleeding
MeSH Terms: conditions — Periodontitis; Hemorrhage

STUDY DESIGN:
Intervention Model Description: an open-label, single-arm clinical study comparing pre- and post-treatment effects
Masking Description: an open-label, single-arm clinical study comparing pre- and post-treatment effects
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 35kDa hyaluronan fragment HA35 injection (Experimental): The investigator injected 35kDa hyaluronan fragment HA35 into the periodontal pocket in a single dose of 100 mg.The distribution of injection amount was determined by the location of gingival inflammation.
  Interventions: Drug: HA35(L20200708MP07707, Ministry of Health, Mongolia) was freshly manufactured by mixing hyaluronidase PH20 injectable solution (H31022111) and high-molecular-weight HA injectable solution (H20174089)

INTERVENTIONS:
Drug: HA35(L20200708MP07707, Ministry of Health, Mongolia) was freshly manufactured by mixing hyaluronidase PH20 injectable solution (H31022111) and high-molecular-weight HA injectable solution (H20174089) — The clinical effects of gingival discomfort oritching, redness and swelling, and bleeding from the probing were observed and recorded in patients before and after 7 days of treatment.
  Other Names: HA35

SUMMARY:
The main objective of this study is to research the treatment of 35 kDa hyaluronan fragment HA35 for Mild periodontitis and associated with gingival discomfort or itchiness.

DETAILED DESCRIPTION:
In this study, tissue permeable 35 kDa low molecular hyaluronan fragment HA35 was freshly manufactured using pharmaceutical grade hyaluronidase PH20 injection (State Drug Administration H31022111) and joint cavity HA injection (State Drug Administration H20174089) mixed at room temperature for 20 min.

In this study, 20 patients, 8 males, and 12 females, with a mean age of 47±15 years, were selected from the outpatient clinic of the Department of Dentistry. All had mild periodontitis and were associated with gingival discomfort or itchiness. Injection treatment was performed using freshly manufactured 35 kDa hyaluronan fragment HA35. The study was an open-label clinical trial in which no information was withheld from the participating investigators. A pre- and post-treatment controlled study approach was used, whereby the investigator injected 35kDa hyaluronan fragment HA35 into the periodontal pocket in a single dose of 100 mg. The distribution of injection amount was determined by the location of gingival inflammation. The clinical effects of gingival discomfort or itching, redness and swelling, and bleeding from the probing were observed and recorded in patients before and after 7 days of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Mild periodontitis and associated with gingival discomfort or itchiness.
2. Patient > 18 years old.
3. Systemically healthy individuals

Exclusion Criteria:

1. Patients who take Anticoagulants or Antiplatelet Agents
2. Pregnant or breastfeeding women
3. Patient having expressed his opposition to participate in the research.

Ages: 32 Years to 62 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-02-02 (Actual); Primary Completion 2023-07-20 (Actual); Study Completion 2023-08-11 (Actual)

PRIMARY OUTCOMES:
Gingival discomfort scores | 7 days
  This study used a modified pain scale to assess gingival discomfort or itching relief. This quantitative assessment represents the degrees of relief of gingival discomfort. Each patient rated their gingival discomfort or itching on a scale of 0 to 10. 0 means "no gingival discomfort or itching" and 10 means "worst gingival discomfort or itching". Pain intensity levels were assessed before and after 7 days of treatment.

SECONDARY OUTCOMES:
The scores of reduction in the extent of gingival redness and swelling and the reduction in gingival bleeding. | 7 days
  Measurement of gum redness and swelling The physician used the numbers 0-10 to rate the intensity of gingival redness and swelling in the subject. 0 means "no gingival redness and swelling"; 10 means "highest intensity of gingival redness and swelling", which is the state of gingival redness and swelling before treatment.
The scores of reduction in gingival bleeding. | 7 days
  Measurement of probe gingival bleeding The physician used the numbers 0-10 to rate the extent to which the subject's probe gums were bleeding. 0 indicating "no gingival bleeding" and 10 indicating "most gingival bleeding from the probe", which is the pre-treatment state.

CONTACTS AND LOCATIONS:
Locations (1):
- Huinuode Biotechnology Co., Ltd., Qingdao, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] APPLICATION OF LOW-MOLECULAR-WEIGHT HYALURONIC ACID(LMW-HA) FRAGMENTS(INJECTION) WO/2017/186088 US20200254005 EP3479830 AU2017255833 CA3049286
- [Result] Jia X, Shi M, Wang Q, Hui J, Shofaro JH, Erkhembayar R, Hui M, Gao C, Gantumur MA. Anti-Inflammatory Effects of the 35kDa Hyaluronic Acid Fragment (B-HA/HA35). J Inflamm Res. 2023 Jan 13;16:209-224. doi: 10.2147/JIR.S393495. eCollection 2023. PMID 36686276
- See also: Related Info — http://patentscope.wipo.int/search/en/detail.jsf?docId=CA249072967&_cid=P22-LDWT33-38680-1DescriptionRelatedInfo